CLINICAL TRIAL: NCT06305039
Title: Optimizing Bilateral and Single-sided-deafness Cochlear Implants for Functioning in Complex Auditory Environments - Part 2
Brief Title: Optimizing Bilateral and Single-sided-deafness Cochlear Implants for Functioning in Complex Auditory Environments
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Walter Reed National Military Medical Center (U.S. Federal Agency); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Matthew Goupell, Professor, Department of Hearing and Speech Sciences, University of Maryland, College Park
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2089705; 1R01DC020506-01A1 (NIH)
Record Dates: First submitted 2024-02-16; First posted 2024-03-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural; Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Bilateral Cochlear Implant Users (Experimental)
  Interventions: Diagnostic Test: Diagnostic tests of cochlear implant or acoustic hearing function; Behavioral: Targeted aural rehabilitation of the poorer performing ear
- Unilateral Cochlear Implant Users with Single-Sided Deafness (Experimental)
  Interventions: Diagnostic Test: Diagnostic tests of cochlear implant or acoustic hearing function; Behavioral: Targeted aural rehabilitation of the poorer performing ear
- Non-Implanted Listeners with Acoustic Hearing (Other)
  Interventions: Diagnostic Test: Diagnostic tests of cochlear implant or acoustic hearing function

INTERVENTIONS:
Diagnostic Test: Diagnostic tests of cochlear implant or acoustic hearing function — Because the cochlear implant participants in the study will use cochlear implant devices that they have already received as part of their standard-of-care treatment, the medical device itself is not an intervention for the purposes of this study. The intervention here will be to carry out diagnostic tests of cochlear implant or acoustic hearing function. This will include perceptual tests of sound localization, speech understanding in noise, binaural fusion, and loudness comparisons.
Behavioral: Targeted aural rehabilitation of the poorer performing ear — Subjects will undergo listening practice on a tablet computer over headphones at home. For the test group, the aural rehabilitation will be targeted at the poorer ear. For the comparison control group, a sham aural rehabilitation will present speech to both ears.
  Arms: Bilateral Cochlear Implant Users; Unilateral Cochlear Implant Users with Single-Sided Deafness

SUMMARY:
Cochlear implants (CIs) are devices that partially restore hearing for people with severe to profound hearing loss. This research focuses on CI users who use bilaterally implanted devices (two CIs, one on each side) and also "single-sided deafness" (SSD) CI users who use one CI together with good acoustic hearing in their opposite ear. The goal is to measure and understand the impact of large input asymmetries across the two ears. These asymmetries are common in BI-CI listeners and always present in SSD-CI users. Although most CI listeners benefit from a second source of auditory input, this project measures how these asymmetries limit speech understanding and spatial hearing. The long-term goal is countering or compensating for input asymmetries. Electrophysiological measures are used to describe the health of the auditory system. Behavioral measures are used to assess if training improves performance. CT imaging is utilized to describe the placement of the CIs.

ELIGIBILITY:
For Bilateral Cochlear Implant Users Arm:

Inclusion Criteria:

* two cochlear implants
* acquired their hearing loss during adulthood or late childhood (post-lingual onset)
* native English speaker
* primarily use oral language
* at least six months of cochlear implant use
* Sufficient corrected or uncorrected visual acuity (20/50 or better) to read large-font text

Exclusion Criteria:

* people who do not use oral language will be excluded.
* people with less than six months of device use will be excluded
* other known disability or neurological disorder
* women who are pregnant will be excluded from the CT portion of the study
* people with any unaided audiometric tone-detection threshold better than 60 dB HL at standard audiometric frequencies (250-8000 Hz) in either ear will be excluded

For Unilateral Cochlear Implant User with Single-Sided Deafness Arm:

Inclusion Criteria:

* one cochlear implant in one ear and a second ear with some acoustic hearing
* acquired their hearing loss during adulthood or late childhood (post-lingual onset)
* native English speaker
* primarily use oral language
* at least six months of cochlear implant use
* Sufficient corrected or uncorrected visual acuity (20/50 or better) to read large-font text

Exclusion Criteria:

* people who do not use oral language will be excluded.
* people with less than six months of device use will be excluded
* other known disability or neurological disorder
* women who are pregnant will be excluded from the CT portion of the study
* people with any unaided audiometric tone-detection threshold better than 60 dB HL at standard audiometric frequencies (250-8000 Hz) in the implanted ear will be excluded
* people with an acoustic pure-tone average threshold (octave frequencies 250-4000 Hz) > 30 dB HL in the non-implanted ear

For Non-Implanted Listeners with Acoustic Hearing Arm:

Inclusion Criteria:

* audiometrically normal hearing or near-normal hearing, or mild/moderate hearing loss
* Sufficient corrected or uncorrected visual acuity (20/50 or better) to read large-font text

Exclusion Criteria:

* severe hearing loss
* other known disability or neurological disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Perceptual responses to sound level | Post-treatment - after at least 6 months use of a cochlear implant if CI user. After enrollment for non-implanted listeners with acoustic hearing.
  Interaural loudness mismatch is defined as the difference between the levels required to balance interaural loudness for sequential stimulation and the levels required to perceptually center a sound image in space for simultaneous stimulation. Participants will respond through pressing virtual buttons on a computer screen. Depending on the condition tested, the sounds will be delivered to one or both ears.
Speech understanding in the presence of masking sounds | Post-treatment - after at least 6 months use of a cochlear implant if CI user. After enrollment for non-implanted listeners with acoustic hearing.
  Speech understanding will be assessed as the percentage of correctly identified keywords.
  Subjects will respond through oral report (where the responses will be scored by the experimenter) or through pressing virtual buttons on a computer screen. The speech sounds will be delivered to one or both ears in the presence of different types of masking sounds. In some cases, signal processing techniques will be used to distort the speech signals to simulate asymmetric hearing abilities.
Computed-tomography scan | For CI users: CT scan will be collected from existing medical records with permission or taken after study enrollment. Measurements taken after study enrollment. Not collected for non-implanted listeners with acoustic hearing.
  A computed tomography temporal bone scan will be used to image the cochlear structures and cochlear implant electrode array located within. This scan will use a standard clinical scanner, with software updated to extend the Hounsfield range to reduce artifact from the metal contacts of the electrode array. This procedure uses radiographic processes, and therefore presents the subject with a safe but nonzero amount of radiation. The CT scan will be analyzed to provide measurements of each array's insertion depth within the cochlea (in degrees and mm), the distance to the cochlear modiolus (mm), and cochlear scalar location.
Electrode impedance (transelectrode impedance matrix) | Post-treatment - after at least 6 months use of a cochlear implant if CI user. Not collected for non-implanted listeners with acoustic hearing.
  This standard clinical measurement will apply a current to one electrode, and measure the resulting induced voltage at each of the other electrodes in the array, one at a time. This process uses low-level electrical stimulation only intended to measure the impedance of the intervening tissues and fluids of the cochlea, and is rarely even perceived by the subject.
Electrically evoked compound action potentials (ECAPs) | Post-treatment - after at least 6 months use of a cochlear implant if CI user. Not collected for non-implanted listeners with acoustic hearing.
  Electrically evoked compound action potentials (ECAPs) will be measured using clinically-available software to track the growth in auditory nerve response (observed ~0.2-0.8 ms post-stimulus onset) as input level is varied from threshold to the maximal level at which the signal is comfortably loud. The slope of input-output function will be measured ( in microvolts/current unit) for each electrode along the electrode array of each cochlear implant study participant.

SECONDARY OUTCOMES:
Sound Localization | Post-treatment - after at least 6 months use of a cochlear implant if CI user. After enrollment for non-implanted listeners with acoustic hearing.
  Participants' ability to localize a virtual sound source in space will be measured. Subjects will be presented with a broadband sound, with signal processing applied (temporal delays and spectral shaping) to simulate a spatial location of the sound source. Subjects will respond through pressing virtual buttons on a computer screen.
Perceptual Fusion | Post-treatment - after at least 6 months use of a cochlear implant if CI user. After enrollment for non-implanted listeners with acoustic hearing.
  Participants' ability to perceptually fuse sounds presented to the ears will be measured. Subjects will be presented with a broadband sound, and will respond through pressing virtual buttons on the computer screen as to (1) how many sounds were heard and where they were perceived inside the head, or (2) which of two mixtures presented contained a larger number of voices.
Spectrotemporal ripple sensitivity | Post-treatment - after at least 6 months use of a cochlear implant if CI user. After enrollment for non-implanted listeners with acoustic hearing.
  This test will be used to evaluate asymmetry in a perceptual measure thought to reflect the peripheral contribution to intersubject variability in speech understanding. This will allow for a baseline from which to ask if the electrophysiological measures provide additional predictive power regarding contralateral disruption beyond the perceptual measures of peripheral asymmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Goupell, PhD, Principal Investigator — University of Maryland, College Park; Joshua G. Bernstein, PhD, Principal Investigator — Walter Reed National Military Medical Center; University of Maryland, College Park
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Maryland, College Park, College Park, Maryland

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that document, support, and validate research findings will be made available when the main findings have been accepted for publication. De-identified data relevant to the project will be disseminated to researchers on and off-campus by request and review of the PI.
  After publication, research products from this project will be archived at the Digital Repository at the University of Maryland(DRUM). DRUM is a long-term, open access repository managed and maintained by the University of Maryland Libraries. Researchers and the general public can download data and code files, associated metadata and documentation, and any guidelines for reuse.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication, available for at least seven years.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee